CLINICAL TRIAL: NCT05092139
Title: enDovascular trEatmenT for acutE isChemic sTroke in China (DETECT2-China): a Prospective, National, Multi-center, Registry Study
Brief Title: Endovascular treatmenT for Acute Ischemic Stroke in China (DETECT2-China)
Status: Completed | Type: Observational
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Head of Neurology, General Hospital of Shenyang Military Region
Other Study IDs: y (2021) 077
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: endovascular treatment — all enrolled patients must receive endovascular treatment

SUMMARY:
This is a prospective real world registry study, aiming to explore the effectiveness and safety of endovascular treatment of acute ischemic stroke in a Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18;
* Ischemic stroke confirmed by head CT or MRI;
* Patients receiving endovascular treatment;
* First ever stroke or pre-stroke mRS≤2;
* signed informed consent.

Exclusion Criteria:

* Prestroke mRS≥3;
* Other serious illness that would confound the clinical outcome at 90 days;
* Unavailable neuroimaging data;
* Other unsuitable conditions judged by the investigator

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: acute ischemic stroke with large vessel oclussion
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with modified Rankin Score 0 to 2 | Day 90
  the minimum and maximum values of modified Rankin Score are 0 and 6, respectively; higher score mean a worse outcome

SECONDARY OUTCOMES:
Proportion of patients with modified Rankin Score 0 to 1 | Day 90
  the minimum and maximum values of modified Rankin Score are 0 and 6, respectively; higher score mean a worse outcome
Distribution of modified Rankin Score | Day 90
  the minimum and maximum values of modified Rankin Score are 0 and 6, respectively; higher score mean a worse outcome
Changes in National Institute of Health stroke scale (NIHSS) | 24 hours, 48 hours, and 2 weeks
  the minimum and maximum values of NIHSS are 0 and 24, respectively; higher NIHSS mean a worse outcome
Proportion of symptomatic intracranial hemorrhage (sICH) | 48 hours
  sICH was defined as 4 or more increase in NIHSS caused by hemorrhage
Proportion of death | 7 days
  death due to any cause

OTHER OUTCOMES:
neuroimaging associated with clinical outcome | 48 hours
  neuroimaging included brain CT, MRI or digital subtraction angiography
changes in serum biomarkers | 48 hours
  biomarker included Matrix metalloproteinases, proinflammatory cytokines, and etc.
dynamic changes of TCD data associated | 24 hours
  transcranial Doppler (TCD) data including blood velocity and pulse index, which will be collected at some centers
dynamic changes of cortical blood oxygen saturation by near infrared spectroscopy | 24 hours
  The data will be collected at some centers

CONTACTS AND LOCATIONS:
Locations (1):
- Hui-Sheng Chen, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu L, Nguyen TN, Chen HS. Endovascular Treatment for Acute Ischemic Stroke in China: a study protocol for a prospective, national, multi-center, registry study. Front Neurol. 2023 Aug 10;14:1171718. doi: 10.3389/fneur.2023.1171718. eCollection 2023. PMID 37638196